CLINICAL TRIAL: NCT05606835
Title: The Effect of Different Subtalar Joint Pronation Amounts on Postural Stability and Lower Extremity Alignment in Healthy Individuals
Brief Title: The Effect Subtalar Joint Pronation on Postural Stability and Lower Extremity Alignment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Collaborators: Acibadem University (Other)
Responsible Party: Principal Investigator, Pelin Pişirici, Assistant Professor, PT, PhD, Bahçeşehir University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: LEA-BAU-AU
Record Dates: First submitted 2022-10-31; First posted 2022-11-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Postural Stability; Dynamic Knee Valgus; Injury Prevention
Keywords: Foot posture; Balance; Tibial torsion; Calcaneal valgus; Frontal plan projection angle

STUDY DESIGN:
Intervention Model Description: Participants will be selected from healthy individuals aged 18-40 years. According to the foot posture index, participants who has a value between 6 and 9 will be added to pronation group and participants who has a value between 10 and 12 will be added to hyper pronation group. Then measurement will be done by the same physiotherapist. Only one measurement will be done.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pronation Group (Active Comparator): Participants will be assessed using the foot posture index-6 (FPI-6), and those who exhibit pronation of the subtalar joint will be included in the study. Participants to be included in the study will be divided into two groups according to their values for pronation increase in the subtalar joint. Participants with a value between 6 and 9 according to FPI-6 will be included in pronation group.
  Interventions: Other: Postural stability assessment; Other: Frontal plan prjection angle; Other: Foot and Ankle Ability Measure; Other: Navicular Drop Test; Other: Calcaneotibial Angle Measurement; Other: Tibial Torsion Angle; Other: Femoral internal and external rotation measurement
- Hyper pronation group (Active Comparator): Participants with a value between 10 and 12 according to FPI-6 will be included in hyper pronation group.
  Interventions: Other: Postural stability assessment; Other: Frontal plan prjection angle; Other: Foot and Ankle Ability Measure; Other: Navicular Drop Test; Other: Calcaneotibial Angle Measurement; Other: Tibial Torsion Angle; Other: Femoral internal and external rotation measurement

INTERVENTIONS:
Other: Postural stability assessment — The Biodex Balance System SD (BDS) (Biodex Medical Systems Inc., Shirley, New York, USA) assesses postural stability (PS). Both static PS (SPS) and dynamic PS (DPS) will be assessed. In the DPS assessment, the platform can be tilted 20° in any direction. For static measurement, participants will be asked to stand barefoot on the platform, stand on one leg, keep the knees in 20-30° flexion. Meanwhile the contralateral knee will be asked to keep in 90° flexion, and stabilize their feet until the end of the test. Upon completion of the SPS assessment, the DPS assessment will be performed. The difficulty level of the DPS test will accepted as 4. For both SPS and the DPS assessment, the test consists of 3 trials of 20 seconds each with a 10-second break between trials.
Other: Frontal plan prjection angle — Frontal Plan Projection Angle (FPPA) is calculated as the angle between the thigh segment and the trunk segment based on the postural image, considering the position of the thigh and tibia. The FPPA will be evaluated using the Spark motion Pro™ application (2D). Before measurement, markers will be placed bilaterally at the SIAS, at the midpoint of the femoral condyles, and at the midpoint of the ankle bones. Participants will stand on the floor barefoot and arms crossed over the chest. Subjects will be asked to squat in a controlled manner and perform a 60° knee bend without losing balance before returning to the starting position. Test will be performed by using single leg squat test. The one-legged squat will be performed for 5 seconds at a standard pace with the researcher acting as the counter. Degrees smaller than 165 will be accepted as increase in knee valgus.
Other: Foot and Ankle Ability Measure — The Foot and Ankle Ailability Measure (FAAM) is used to assess the self-reported overall functional level of patients with leg, foot, and ankle musculoskeletal injuries and conditions. It consists of 1) activities of daily living [ADL] and 2) sports [S] and can be scored from 0 to 100%. In the FAAM, there are 29 items that are scored from 0 to 4. There are 21 items related to various functional activities under the subtitle activities of daily living, and 8 items related to various activities related to participation in sports under the subtitle sports. Standardized response options are answered on five-point likert scales ranging from 0 (I cannot) to 4 (no difficulty). Point totals between 0 and 84 for the ADL subtitle and between 0 and 32 for the Sports subtitle are converted to percentage points.
Other: Navicular Drop Test — The navicular drop test (NDT) is a clinical method for assessing the mobility of the medial longitudinal arch (MLA). The extent of navicular subsidence is assessed to determine the flexibility of the MLA and the position of the navicular with and without transfer of body weight. To assess navicular drop, the subtalar joint will be positioned in neutral position and the height of the navicular will be measured in non-weight bearing position. Then the measurement will be repeated in weightbearing position. The height difference between the two measurements in sitting and standing is recorded as the NDT value. Values more than 10mm is accepted as pathological.
Other: Calcaneotibial Angle Measurement — Measurement of the calcaneotibial angle (CTA) is one of the methods used in the evaluation of the foot and ankle. By measuring this angle, it is assessed whether the ankle problems are related to the hindfoot. In the CTA measurement, the angle between the vertical axis of the calcaneus and the longitudinal axis of the achilles tendon is measured in the standing and prone positions, and the differences will be recorded. Values more than 8 degrees is accepted as calcaneal valgus.
Other: Tibial Torsion Angle — Tibial torsion is a rotational deformity which can be measured between the long axis of the tibia and the transmalleolar axes. This measurement can be used to determine the extent to foot malalignment is due to bone torsion. Measurement will be done by a goniometer. Participants will be asked to lie prone and will be positioned with the knee joint in 90° flexion and the ankle joint in a neutral position. Normal alignment is 20 degrees external rotation. Any increase or decrease accepted as pathological.
Other: Femoral internal and external rotation measurement — Accurate assessment of hip joint range of motion (ROM) is an important component in the overall clinical evaluation of lower extremity injuries, particularly those of the hip and groin. The expected hip rotational range of motion for internal rotation (IR) is 45°, and for external rotation (ER) is 0° to 45°. In this study, a smartphone-based inclinometer will be used to measure femoral IR and ER. The inclinometer will be placed vertically so that the top edge is just below the tibial tuberosity and the bottom edge is pointed at the midpoint of the medial and lateral malleoli.

SUMMARY:
The lower extremity consists of sequent columns. The deviation of one segment from its normal alignment in the lower extremity also affects the alignment of the other segments. The alignment of the parts of the foot during weight bearing is called foot posture. Foot posture is divided into neutral, pronation, and supination. Foot posture varies significantly from person to person, and deviations from normal foot posture are associated with lower extremity injuries. Increased or prolonged pronation has been identified as both a risk factor and etiologic factor for increased navicular drop, a lower extremity malalignment pattern. In pronation posture, the foot may not adequately adapt to the ground, and there is increased movement of the lower extremity in the frontal plane. As a result, the person's postural stability is compromised. The fact that the foot is the most distal segment of the lower extremity chain indicates that even small biomechanical changes in the bearing surface can significantly affect postural control strategies. There are studies in the literature that examine the effect of foot pronation on dynamic balance and postural stability in individuals with different foot postures. However, to our knowledge, there is no study that examines differences in postural stabilization and lower extremity alignment by classifying individuals with varying degrees of subtalar joint pronation into pronation and hyper pronation groups.

DETAILED DESCRIPTION:
Examination of the biomechanics of the foot and ankle is an important aspect in the evaluation of human movement. The purpose of this study is to divide healthy subjects into pronation and hyperpronation foot postures and investigate the effects of differences subtalar pronation amounts in lower extremity alignment and postural stabilization. The part of the foot where the subtalar joint is located is called the hindfoot. The anatomy and alignment of the hindfoot is a critical factor in the biomechanics of the lower extremities and the function of human locomotion. Pronation of the foot causes tibial internal rotation and femoral internal rotation through the mechanism of the kinetic chain, resulting in valgus alignment of the knee when the foot is on the ground. The valgus alignment changes the position of the pelvis. Alternations in pelvic position increases the tension on the hip and pelvic muscles because it changes the force lever. In addition, increased femoral internal rotation of the lower extremity relative to the tibia has been shown to increase stress on the weight-bearing tissues of the tibio-femoral compartments and increase tibial internal rotation in individuals with pronated foot posture. Normal pronation motion is necessary for proper foot function, but increased and excessive pronation of the subtalar joint is a condition that should be investigated because it presents several problems with lower extremity alignment. The fact that foot pronation is important for the lower extremity kinetic chain during dynamic tasks prompts us to investigate foot pronation by measuring it in various ways. The purpose of this study is to divide healthy subjects into pronators and hyper pronators and to investigate the effects of differences in lower extremity kinetic chain alignment and postural stabilization and in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18 and 40 years old
* Not to have pain and function loss
* Foot posture index value between 6-12
* No orthopedic disease
* Not be visually or hearing impaired
* Not have participated in a physical therapy program in the past 6 months
* Not have undergone any surgical procedure on the lower extremity
* No intake of pain medication during the examination period and within the specified treatment days

Exclusion Criteria:

* Having congenital anomaly of the lower extremity
* Having a history of lower extremity surgery or lower extremity surgery planned within the next 12 months
* Having ligament hyperlaxity
* Having a history of tendon or cartilage injury
* Having metabolic disease, cancer
* Using any kind of support/orthosis in the shoe
* Having knee injections in the past 3 months
* Any neurological or systemic inflammatory arthritis disorder

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Postural stability assessment | Baseline
  The Biodex Balance System SD (BDS) (Biodex Medical Systems Inc., Shirley, New York, USA) assesses postural stability (PS). Both static PS (SPS) and dynamic PS (DPS) will be assessed on single leg. The investigators will assess postural stability only one time.

SECONDARY OUTCOMES:
Frontal plan prjection angle (FPPA) | Baseline
  2D motion analysis data were evaluated with the Spark Motion Pro™ mobile motion analysis system during the one-leg squat test, a functional test for dynamic knee valgus. FPPAs were measured with the Spark Motion Pro™ goniometry application. The validity and the reliability study of the FPPA measurement in individuals with DDV was conducted by Ramirez et al. in 2018. The use of the application in individuals with DDV was found to be reliable. Degrees smaller than 165 will be accepted as increase in knee valgus. The investigators will assess FPPA only one time.
Foot and Ankle Ability Measure (FAAM) | Baseline
  FAAM is used to assess the self-reported overall functional level of patients with leg, foot, and ankle musculoskeletal injuries and conditions. It consists of 1) activities of daily living [ADL] and 2) sports [S] and can be scored from 0 to 100%. In the FAAM, there are 29 items that are scored from 0 to 4. There are 21 items related to various functional activities under the subtitle activities of daily living, and 8 items related to various activities related to participation in sports under the subtitle sports. Standardized response options are answered on five-point likert scales ranging from 0 (I cannot) to 4 (no difficulty). Point totals between 0 and 84 for the ADL subtitle and between 0 and 32 for the Sports subtitle are converted to percentage points. The investigators will assess FAAM only one time.
Navicular Drop Test (NDT) | Baseline
  NDT is a clinical method for assessing the mobility of the medial longitudinal arch (MLA). The height difference between the two measurements in weight bearing and nonweight bearing is recorded as the NDT value. Values more than 10mm is accepted as pathological. The investigators will assess NDT only one time.
Calcaneotibial Angle Measurement (CAM) | Baseline
  In the CTA measurement, the angle between the vertical axis of the calcaneus and the longitudinal axis of the achilles tendon is measured in the standing and prone positions, and the differences will be recorded. Values more than 8 degrees is accepted as calcaneal valgus. The investigators will assess CAM only one time.
Tibial Torsion Angle (TTA) | Baseline
  TTA Measurement will be done by a goniometer. Participants will be asked to lie prone and will be positioned with the knee joint in 90° flexion and the ankle joint in a neutral position. Normal alignment is 20 degrees external rotation. Any increase or decrease accepted as pathological.
Femoral internal and external rotation measurement | Baseline
  The expected hip rotational range of motion for internal rotation (IR) is 45°, and for external rotation (ER) is 0° to 45°. In this study, a smartphone-based inclinometer will be used to measure femoral IR and ER in sitting position.

CONTACTS AND LOCATIONS:
Overall Officials: Pelin Pişirici, PhD, PT, Study Chair — Bahçeşehir University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation; Özlem Karakaş Fevzioğlu, PhD, PT, Study Director — Acibadem University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation; Gülsüm Bayıroğlu, PT, Principal Investigator — Bahçeşehir University, Graduate Education Institute, Physical Therapy and Rehabilitation Program
Locations (1):
- Pelin Pişirici, Istanbul, Besiktas/Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No